CLINICAL TRIAL: NCT01830634
Title: Effect of Strength and Flexibility Training With Elastic Band on Gait Pattern and Functional Ability in the Elderly
Brief Title: Lower-limb Strength and Flexibility Program on Prevention of Falls in the Community-dwelling Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I050507; NSC-93-2314-B-371-002 (Other: National Science Council)
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Accidental Falls
Keywords: Community-dwelling elderly; Rehabilitation; Theraband; Strengthening and stretching exercise

ARMS (1):
- Theraband with strengthening and stretching exercise (Experimental): All subjects were received theraband exercises (strengthening and stretching), and then compare the measured outcomes between groups.
  Interventions: Behavioral: Theraband with strengthening and stretching exercise

INTERVENTIONS:
Behavioral: Theraband with strengthening and stretching exercise — Using the theraband for strengthening and stretching the upper and lower extremity muscles.
  All exercises were performed by using a Theraband in the following movements: shoulder elevating and abducting, horizontal and oblique direction, plantar flexion, dorsi-flexion, inversion and eversion of ankle, knee extension and hip abduction. The stretching exercises were focused on the hamstring muscle and heel cord. Each movement was held for 5 seconds. The participants were instructed to perform 5-10 repetitions of each movements twice per day.

SUMMARY:
Accidental falls result in major physical and psychological morbidity in the elderly. The aim of this study was to evaluate the effects of lower-limb strength and flexibility program, which is analyzed under the control of other risk factors, on preventing falls and fall-related injuries in the community-dwelling elderly.

DETAILED DESCRIPTION:
To estimate the effect of strength and flexibility training with elastic band on community-dwelling elderly gait, balance, and functional performance. All subjects received a home exercise program with low resistance elastic band training. All subjects were assessed for functional assessment, balance and gait analysis at initial and after training.

ELIGIBILITY:
Inclusion Criteria:

* elder living in community
* age > 65 years old

Exclusion Criteria:

* no walking ability before fall
* conscious change or disease induce fall
* impaired cognition

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2005-06; Primary Completion 2006-01 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Computerized balance evaluation | after 3 months intervention
  computerized balance and gait evaluation by a posturography and gait analysis system

SECONDARY OUTCOMES:
improve in functional activity | after 3 months intervention
  functional reach and timed up-and-go test

CONTACTS AND LOCATIONS:
Overall Officials: TaSen Wei, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital Taiwan, Changhua, Taiwan